CLINICAL TRIAL: NCT02840864
Title: Comparison of Sonographically Assisted With Conventionally Breast Surgery - Prospective, Randomised, Multicenter, Parallel Group Study With Two Study Arms
Brief Title: Comparison of Conventional With Sonography Assisted Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAC-002
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2024-07-22 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Sonographically assisted breast surgery
  Interventions: Device: Sonography assisted breast surgery
- Arm 2 (Active Comparator): Conventional breast surgery
  Interventions: Device: Sonography assisted breast surgery

INTERVENTIONS:
Device: Sonography assisted breast surgery

SUMMARY:
Aim of the study is to test whether surgical removal of a tumor under sonographic control as compared to conventional method reduces the rate of resections and local relapse

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years
* Female
* Presurgical validated breast cancer

Exclusion Criteria:

* Sonographically not defined report
* Lobular breast cancer
* Extensive ductal carcinoma in situ

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2015-07; Primary Completion 2018-04 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Rate of second tumor resections | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Women's Health, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No